

# FAPO-X: Assisted digital telemonitoring with wearables in patients after cardiovascular surgery – a randomized trial

financed by samsung

Researchers: Prof. MD, PhD Fabio Biscegli Jatene
Prof. MD, PhD Carlos Alberto Pastore
Prof. PhD Marco Antonio Gutierrez
Eng. Fabio Pires
BSc, Phd, Rosangela Monteiro
Eng. Guilherme Rabello
BSc, PhD Camila Rodrigues Moreno
Pietro Colonna
Nurse, MSc. Matheus Moitinho
Nurse Bruna Lopes

Sao Paulo January 07, 2023







#### **SUMMARY**

| | | | Page |
|---|---|---|---|
| 1 | INTR | ODUCTION | 1 |
| 2 | GOA | LS | 9 |
| | 2.1 | goal primary | 9 |
| | 2.2 | Goals secondary | 9 |
| 3 | METH | HODOLOGY | 9 |
| | 3.1 | Study location | 9 |
| | 3.2 | Inclusion criteria _ | 10 |
| | 3.3 | Exclusion criteria _ | 10 |
| | 3.4 | Selection of Volunteers | 10 |
| | 3.5 | Data collection, clinical examinations and evaluation of results | 13 |
| | 3.6 | Validation of the Measurement Model and Data Analysis | 15 |
| | 3.7 | Anamnesis complete | 15 |
| | 3.8 | Provision and use of SAMSUNG devices (smartphone | 16 |
| | | and smartwatch ) | |
| | 3.8 | Traditional electrocardiography (ECG) versus | 16 |
| | | SAMSUNG smartwatch ECG | |
| | 3.9 | Measurement of peripheral oxygen saturation (SpO2) by | 17 |
| | | SAMSUNG smartwatch versus standard oximetry | |
| | 3.10 | Blood pressure (BP) measurement by SAMSUNG | 17 |
| | | smartwatch versus standard device | |
| | 3.11. | Definition of alerts - teleassisted group | 18 |
| | 3.13. | Aspects ethical | 23 |
| | 4. | Timeline Estimated | 24 |
| | 5. | Attachments | 25 |
| | 5.1. | case report Form (CRF) | 25 |
| | 5.2. | Term of Loan Liability | 33 |
| | 5.3 | Activity Diary | 35 |
| | | References | 37 |





#### 1. INTRODUCTION

Noncommunicable diseases are responsible for about 41 million deaths/year, which is equivalent to 71% of deaths worldwide <sup>1</sup>. It is no different in Brazil, chronic diseases represent the main challenge in health, about 72% of deaths in the country are due to chronic non-communicable diseases, which represent 75% of the expenses of the Unified Health System (SUS) - Figure 1.



Figure 1. Chronic diseases represent the main health challenge in Brazil.

The World Health Organization's 2030 Agenda for Sustainable Development reveals the commitment of member countries to a 30% reduction in premature mortality from non-communicable diseases, especially cardiovascular diseases (ischemic heart disease and stroke), cancer, respiratory disease and diabetes <sup>2</sup>.







Cardiovascular diseases represent one of the major causes of morbidity and mortality worldwide, which has encouraged numerous researches in different areas. Around 17.5 million people die from cardiovascular diseases annually worldwide, according to data from the World Health Organization (Figure 2). Only in Brazil, diseases related to heart problems correspond to about 300,000 deaths per year. They are chronic and can be treated clinically or surgically <sup>3</sup>.

Figure 2 . Leading causes of death worldwide in the year 2019.



A significant portion of cardiovascular diseases require surgical treatments, with myocardial revascularization surgeries, correction of valve diseases, followed by surgeries to correct aortic diseases and congenital heart diseases, the most common in adults and the elderly. These patients are usually referred to the operating room with different comorbidities, subject to more complications in the







intra and postoperative period, which leads to an increase in hospital stay and monetary and technological costs invested in their treatment and recovery <sup>4, 5</sup>.

Brazil is the second country in the world in number of heart surgeries performed, totaling around 100,000 surgeries/year, second only to the USA, which performs around 300,000 surgeries/year.

There are over 320 million inpatient surgical procedures performed worldwide. Recently, the *International Surgical Outcomes (ISOS) Study (ISOS Group 2016)* highlighted that about 17% of these patients develop one or more complications and, among them, 2.8% die as a result of them <sup>6, 7</sup>.

The postoperative period of cardiac surgery requires continuous observation from the health team, quick decision-making and highly complex care. This period presents many challenges for the multidisciplinary team, due to the need for intensive/constant monitoring and the potential postoperative complications. In addition to the lives lost, these postoperative complications dramatically increase hospital and healthcare costs <sup>8</sup>.

One of the most frequent complications in the postoperative period of cardiovascular surgery are arrhythmias, with atrial fibrillation being the most frequent arrhythmia in the postoperative period <sup>9</sup>. The prevalence of postoperative atrial fibrillation (POAF) varies between 15 and 40% in coronary artery bypass grafting procedures, 37 to 60% in valve surgery and more than 60% in combined interventions and 24% in patients undergoing heart transplantation.

In 90% of cases, POAF appears in the first four postoperative days <sup>10</sup>. The average length of the first episode is 7-8 hours. Recurrence occurs in 40% of cases and occurs within the first 24 hours. Up to 80% of patients remain in sinus rhythm







24 hours after the first episode. About 14% of patients with atrial fibrillation after cardiac surgery (AFACS) remain with this rhythmic disorder for up to two weeks <sup>11</sup>.

Other emerging evidence suggests that POAF is associated with long-term sequelae such as stroke, heart failure, and all-cause <sup>12</sup>mortality. <sup>13</sup>

Despite the advances in the area and the different methods for monitoring POAF, there is still no method that allows the automated evaluation of fibrillation episodes for a very prolonged period. Thus, the detection of POAF becomes an important challenge.

Wearable devices such as *smartphones* and *smartwatches*, are a great promise for screening and monitoring AF, and can present up to 93% sensitivity and 84% specificity when compared to standard ECG <sup>14</sup>. In addition, they are easy to use and allow evaluating the possible adherence of patients to this new modality of assisted telemonitoring. However, to be used as a medical device, these *wearables* need to be accurate in outpatient settings.

#### Technological resources for health solution

The use of terms such as Internet of Things or *Internet of Things* ( IoT ), Internet of Everything or *Internet of Everything* ( IoE ), cloud computing, cyberculture, big data, artificial intelligence, neural networks, wearable devices, among *others*, are already part of our daily lives as innovative technological contributions in the area of health <sup>15, 16</sup>.

Wearables are proving to be very effective tools with regard to the prevention, detection or even management of chronic diseases, according to Baig et al <sup>17</sup>. The use of *wearables* to monitor vital signs, such as oxygen saturation (SpO2), heart rate, blood pressure and respiratory rate is of fundamental







importance <sup>18</sup>. In addition, the possibility of generating early warnings in case of clinical instability of the patient was associated with a significant decrease in the number of cardiac arrests and deaths <sup>19</sup>. Statistical data and trend models, even generated from non-medical devices such as *wearables*, are of great value in preventive and predictive actions in health care <sup>20</sup>, <sup>21</sup>.

The use and implementation of any new technology comes at a cost that must be balanced against the potential savings associated with the expected improvement in postoperative recovery. Postoperative complications are expensive to treat and prolong hospital stays. However, the use of such resources as *wearables* will allow a variety of data to be collected by sensors and allow for earlier interventions <sup>22</sup>.

Recent data from a GFK36 global survey on *wearables*, involving more than 20,000 people in 16 countries, found that around 33% use tracking to monitor their health, through apps, bracelets, smart watches and clips. Among those interviewed, 18% had already used the technology some time ago, 45% had never used it and 4% were unable to answer. This survey revealed an interest in wellness, looking for information about exercise, calorie consumption, and even sleep. Another interesting data from this survey is that Brazil occupies, alongside the United States, the second position in the use of health and physical condition monitoring, losing to China and ahead of Germany and France <sup>23</sup>.

In this context, the use of available technologies can be used as strategies for faster dehospitalization, with remote monitoring of the patient, since the initial application of *wearables* in surgery may eventually allow better communication and decision-making by the care team through the collection, interpretation and







presentation of patient-specific measurements relevant to the context of the disease <sup>24</sup>.

Wearable devices, such as smartwatches, can be an innovative and relevant alternative, making it possible to reduce hospitalization periods and the early return of patients to their routine activities safely, in an assisted way.

#### Integration of wearable technology health data with the electronic record

Currently, Information and Communication Technology (ICT) tools are present in practically all activities related to the health area, such as teaching, research or assistance.

There is evidence that a feasible and adequate electronic health record (EHR) helps professionals in decision-making in patient health care, improving safety and efficiency of care <sup>25</sup>. In view of this, there has been a progressive interest in the medical field in using data captured from the RES, as they contain variables with valuable information, such as demographic data, diagnoses, medications and laboratory data <sup>26, 27</sup>.

However, although electronic records serve different purposes and utilize different IT system architectures, there are many operational challenges and technical issues. However, the different needs and subdivisions of the health area, without a systematic view, end up using an exaggerated amount of software and spreadsheets, without interconnection or integration, making it difficult or even preventing the communication and transformation of data into relevant information and knowledge in practice. clinic <sup>28</sup>, <sup>29</sup>.

InCor's electronic medical record (Integrated Information System InCor - SI<sup>3</sup>) provides integrated data from the Clinical Information System via a standard web







interface, which allows independence from the hardware platform *used* for access, in addition to providing better management of health resources in the institution, whether in supplies, occupation of beds, laboratory management, medications, costs of procedures and information that can be obtained in real-time through standardized interfaces <sup>30</sup>. Currently, more than 1.4 million patients are registered in SI3 with all their care data, resulting in more than 500 Terabytes of data. The systems range from scheduling appointments and exams and admitting patients to bed control, laboratory management, medication, supplies and billing to the SUS.

In this way, not only the secure integration of the currently existing databases, but also the coherent use of the stored information, provide a valuable source of knowledge for a better understanding of patients treated by the SUS, thus allowing exploratory, prospective and retrospective studies to produce predictive models, and facilitating decision-making for better management of public health policies.

Wearable technology, such as the use of *smartwatches*, can capture valuable bioparameters, and that at the same time, EHR provides practical platforms for including these data - the creation of a graphical interface that displays patients' health data from these devices could both transform medical care and ensure patient privacy.

In view of the above, the present study aims, through the use of the **Smartwatch SAMSUNG** <sup>TM</sup> **Galaxy Watch5**, to validate a measurement model and data analysis that early indicate the need for medical assistance due to atrial fibrillation (AF) in individuals with heart disease undergoing cardiac surgery, as well as to evaluate patients' commitment to a new monitoring routine using regular







alerts based on automated readings, in comparison with the traditional postoperative routine.

The use of such devices as predictors of cardiac alterations could save the SUS hundreds of millions of reais per year, as it would avoid events in these individuals and, consequently, their treatment. To this end, this study will be randomized so that 50 patients will use a *Smartwatch device SAMSUNG* TM *Galaxy Watch5* and 50 patients will follow the institution's standard treatment (not monitored by wearables).

#### 2. OBJECTIVES

#### 2.1 Primary Purpose

telemonitoring platform using the *Smartwatch SAMSUNG ™ Galaxy Watch5*, validating its applicability in patients with POAF.

#### 2.2 Secondary objectives

- Evaluate the accuracy of the Smartwatch SAMSUNG ™ Galaxy Watch5
  in detecting vital signs through optical sensors and, in particular, possible
  heart rhythm irregularities.
- Compare the results of the variables heart rate, blood pressure and peripheral oxygen saturation (SpO₂) and electrocardiogram provided by the 
  \*\*Smartwatch SAMSUNG \*\* Galaxy Watch5\* with data obtained from gold standard reference equipment.





#### 3. METHODOLOGY

#### 3.1 Place of study

This project will be carried out entirely on the premises of the Instituto do Coração of the Hospital das Clínicas of the Faculty of Medicine of the University of São Paulo. The sample will consist of 100 outpatients, with heart disease undergoing cardiac surgery, and selected during the pre -surgical consultation. The sample size was proposed by the contractor because it is a pilot study to evaluate the accuracy of the equipment in a sample with POAF.

#### 3.2 Inclusion criteria

- Be at least 22 years old;
- Parameters for surgical indication, in the presence of heart disease (mitral or aortic valve disease, coronary artery disease or aortic disease);
  - Agree to adhere to the study's procedures and requirements;
  - Be able to consent to their participation in writing;
  - Possess home internet connectivity infrastructure;

#### 3.3 Exclusion criteria

- Not having undergone cardiac surgery;
- Presence of post-surgical complications with prolonged hospital stay for more than 14 days from surgery date;
- Presence of a Peripherally Inserted Central Catheter (PICC) or limb preservation and cardiac pacemaker in case of impediment to acquisition of the ECG (smartwatch);
- Patients with arteriovenous fistula;
- Presence of skin pathology or skin diseases such as vitiligo, lupus and atopic dermatitis, as well as tattoos in the wrist region, which may interfere with the reading by the optical sensor;
- Show sensitivity or allergic reactions, to any degree, to the component materials of the wearable device:







Volunteers who meet the research inclusion criteria will participate in the study protocols after signing the informed consent form (TCLE).

#### 3.4 Selection of volunteers

Patients with heart disease undergoing cardiac surgery, monitored at the InCor outpatient clinic. Randomization will be performed 1:1 using an electronic randomization system and subsequently stratified from the RedCap platform, without knowledge by the team involved in the study. Patients will be randomized to intervention group (teleassisted group) or control group (standard follow-up of the institution)

- Control group (N=50): patients with heart disease who underwent a surgical procedure with standard outpatient and post-surgical follow-up, according to institutional routines and protocols;
- Tele-assisted group (N=50): patients with heart disease undergoing a surgical procedure remotely monitored through smartwatch and application.

Adult patients will be included, of both sexes, and ethnic profile representative of the Brazilian population, characteristic of the user population of the Unified Health System (SUS).

re-hospitalization rate, through scheduled consultations and extra intercurrences (clock x institutional standard). As secondary outcomes will be evaluated: technological and treatment adherence, through the use of the mobile application by patients and development and implementation of the telemonitoring platform.

The goal is the inclusion of 40 patients/month (in all, in the 2 study groups: Remotely monitored watch group and group without a watch, following the institutional standard, following the randomization order generated by a specific



system) with 20 in each group of the study. In addition, the inclusion of patients will happen gradually and continuously, with 1 patient per group/working day.

| Sem 1 Sem 2 Sem 3 | | Sem 4 Sem | | Sem 6 | Sem 7 | Sem 8 | Sem 9 | |
|---|---|---|---|---|---|---|---|---|
| 1 ao 5 | 6 ao 10 11 ao 15 | | 16 ao 20 | 21 ao 25 26 ao 30 | | 31 ao 35 | 36 ao 40 | 41 ao 45 |
| | | | | | | 1 ao 3 | 4 ao 8 | 9 ao 13 |
| Sem 10 | Sem 11 | Sem 12 | Sem 13 | Sem 14 | Sem 15 | Sem 16 | Sem 17 | |
| 46 ao 50 | | | | | | | | |
| 14 ao 18 | 19 ao 23 | 24 ao 28 | 29 ao 33 | 34 ao 38 | 39 ao 43 | 44 ao 48 | 49 ao 50 | |
| <ul> <li>Inclusão ● Retorno</li> </ul> | | | | | | | | |

Figure 3. Flow of inclusion of patients in each arm of the study.

The remote patient monitoring flowchart to be used in this project is shown in Figure 3. Briefly, it includes:

- 1. Preoperative outpatient consultation with complete anamnesis to verify eligibility for using the SAMSUNG \*\*M\*\* Galaxy Watch5 Smartwatch;
- 2. Hospitalization, surgery and collection of intraoperative data;
- Training of the patient and/or family member responsible for the use of smartwatch and smartphone to start post-operative remote monitoring;
- 4. Upon hospital discharge, the patient will receive guidance for follow-up on the platform with the *Smartwatch SAMSUNG <sup>TM</sup> Galaxy Watch5*;
- 5. Remote patient monitoring with **SAMSUNG** TM **Galaxy Watch5 Smartwatch** and app for 30 ± 3 days;
- 6. Monitoring by InCor's multidisciplinary team of the parameters collected using the Smartwatch SAMSUNG ™ Galaxy Watch5 and an application installed on a smartphone; identifying risks for early interventions in the face of any relevant intercurrence;





- 7. Remote monitoring of the patient by teleconsultation, in case of detection of intercurrences. In cases considered serious by the clinical team, patients will be instructed to seek the InCor PS;
- 8. Face-to-face return to the outpatient clinic  $30 \pm 3$  days after discharge for evaluation by the clinical team and conclusion of participation in the study.



Figure 4. Proposed flowchart for the project.

#### 3.5 Data collection, clinical examinations and evaluation of results

In this project, wearable devices such as the Galaxy Watch will be used. 5 together with Galaxy series smartphones (A or S line) for the acquisition of blood pressure measurements, arterial hemoglobin oxygen saturation (SpO2), heart rate and ECG. This data will be transmitted to a repository, in a secure cloud environment, which meets the requirements of the General Data Protection Act





(LGPD) (Figure 5). In addition, data will be transmitted to a platform to be developed by InCor's IT team, as part of the project, and integrated into InCor's electronic medical record through the WebAdmin tool.



Figure 5 . Conceptual diagram for the Telemonitoring Platform.

The division of the study into phases and activities was carried out according to the table and description below.

| Phase | Local | Activity |
|---|---|---|
| Phase 1 | outpatient | <ul> <li>Inclusion of patients</li> <li>Preoperative consultation;</li> <li>Meeting with the project coordination team;</li> <li>Complete anamnesis;</li> <li>Application of the TCLE;</li> <li>Collection of additional and contact information;</li> </ul> |
| Level 2 | hospitalizati<br>on | <ul> <li>Hospitalization;</li> <li>Eventually, some patients may be included in the study after hospitalization, prior to surgery, with the application of informed consent at this time;</li> </ul> |
| phase 3 | surgical | <ul> <li>Performing the surgical procedure;</li> <li>Intraoperative data collection;</li> <li>Postoperative evaluation and discharge</li> <li>Patient guidelines;</li> <li>Signature of the equipment loan liability term (smartphone and smartwatch); and the term for using data from the Electronic Health Record;</li> <li>Calibration:</li> <li>BP, serial measurements - smartwatch SAMSUNG + traditional auscultatory method;</li> <li>ECG - smartwatch SAMSUNG + traditional ECG;</li> <li>SpO2 - SAMSUNG smartwatch oximetry + traditional oximetry;</li> <li>Questionnaire of events observed during the remote phase;</li> </ul> |





| Phase 4 | remote<br>collection | <ul> <li>Tracking, monitoring and managing each participant's remote data collection for 30 ± 3 days; these being: <ul> <li>Automatically collected: SpO2, heart rate, steps and sleep.</li> </ul> </li> <li>Collected manually: blood pressure and ECG.</li> <li>Telephone contact, teleconsultations, and unscheduled face-to-face consultations in cases of complications;</li> </ul> |
|---|---|---|
| Phase 5 | outpatient | <ul> <li>Return outpatient consultation;</li> <li>Meeting with the project coordination team;</li> <li>Return of equipment used in the remote phase;</li> <li>ECG - smartwatch SAMSUNG;</li> <li>SpO2 - smartwatch SAMSUNG + traditional oximetry;</li> <li>PA - smartwatch SAMSUNG + traditional auscultatory method;</li> <li>Quality of life questionnaire adapted to record the patient's perception during the remote monitoring phase;</li> <li>Issuance of a report confirming or not the classification of the ECG issued by the smartwatch;</li> </ul> |
| phase 6 | InCor | <ul> <li>Description of tests carried out and compilation of final results;</li> <li>Definition, description and justification of the statistical tests chosen and aligned with the hypotheses raised at the beginning of the study.</li> </ul> |

Table 1: Protocol phases, locations and activities.

#### 3.6. Validation of the Measurement Model and Data Analysis

The measurement validity of *wearables* will be checked against standard reference methods used at InCor, in order to verify the effectiveness of using *wearables* using parametric or non-parametric statistical tests, depending on the normality distribution pattern of the variables to be studied, considering p values <0.05 statistically significant.

The identification, sociodemographic and clinical data of the patients will be registered in the REDCap program, considered as a tool for managing and storing research data<sup>31</sup> and analyzed using *Statistical Package for the Social Sciences* (SPSS) version 22.0 for Windows.

#### 3.7 Complete anamnesis

After confirming participation in the study, initial clinical examinations should be scheduled. Volunteers will be assessed for family and personal health history, and the variables to be collected are described in the case report Form (CRF) of the study (Annex 2).





## 3.8 Provision and use of SAMSUNG devices (smartphone and smartwatch)

**SAMSUNG** devices will need to be handed over to participants in phase 3 of the study in order for remote data collection to begin. Volunteers must sign a loan liability term that guarantees the return of the device, and coverage in case of damage, as per Annex 3. Longitudinal data collection will be carried out for a period of 30 days ± 3 days, requiring remote monitoring by team. Smartphones and *smartwatches* will be used to monitor adverse events regarding cardiac arrhythmia, heart rate *and* blood pressure. All devices will be delivered with the necessary applications for data collection duly installed. However, customization (login and initial settings) will be carried out by the Innovation team. During phase 4, each participant will remain with **SAMSUNG** devices for 30 days ± 3 consecutive days. Participants must use the *smartwatch* and *smartphone* throughout the day, including while sleeping, and charge the equipment batteries regularly. The data will be collected by an application embedded in the equipment.

During phase 5, the participant must return to InCor for a final consultation of the study, and return of borrowed equipment.

## 3.8 Traditional electrocardiography (ECG) versus SAMSUNG smartwatch ECG

Still in phase 3 of the project, resting electrocardiography (ECG) tests will be performed in conjunction with ECG collection from the *smartwatch* **SAMSUNG**, for comparison between the two analysis methods (gold standard vs. device).

All electrocardiograms will be performed at a speed of 25mm/ sec, with 1mV/10mm calibration, in a MAC 2000 ECG Machine (GE Medical Systems Information Technologies, Inc., WI, USA) on an outpatient basis. The electrodes will be placed in the classic way of 12 leads (6 in the frontal plane D 1,D 2,D3,aVr,aVl,aVf and 6 in the horizontal plane V1,V2,V3.V4,V5,V6 ). The parameters will be evaluated by the clinical cardiologist, who will issue a report, based on the guidelines of the Brazilian Society of Cardiology on analysis and issuance of electrocardiographic reports.





## 3.9 Peripheral oxygen saturation (SpO<sub>2</sub>) measurement by SAMSUNG *martwatch versus* standard oximetry

SpO<sub>2</sub> values will be measured simultaneously by the *smartwatch* **SAMSUNG** and a digital pulse oximetry equipment (G-TECH 302L). Traditional oximetry, using an infrared light beam, simultaneously measures heart rate and peripheral oxygenation in percentages of 0-100%, and measurements above 95% will be considered normal. This evaluation will be carried out in phases 3 and 5 of the project.

## 3.10 Blood pressure (BP) measurement by SAMSUNG *smartwatch* versus standard device

smartwatch will first be calibrated **SAMSUNG** for BP measurement following the instructions of the equipment itself. From then on, 8 consecutive measurements will be taken, at rest, alternating between using the *smartwatch* **SAMSUNG** and the arm pressure gauge (Brand *Welch*) standard, which uses aneroid meter and pulse auscultation (stethoscope *littman clinic*). Measurements with the standard device will be performed with the patient in the supine position, after 10 minutes of rest with 3 consecutive measurements. Additionally, a measurement will be performed in a sitting position and another measurement in an orthostatic position with a 30-second difference between measurements.

This assessment will be repeated in phase 5 of the project, following the same methodology described above.





#### 3. 11 Definition of alerts – teleassisted group

The multidisciplinary team will receive alerts through the application platform, according to pre-established limits of blood pressure, heart rate and blood oxygen saturation.

#### • Blood pressure

Normal Parameters: Systolic [100 – 140 mmHg] and diastolic [70-90 mmHg]

Yellow Alert: Systolic [100 – 180 mmHg] and diastolic [90 – 110 mmHg]

Red Alert: Systolic [<90 and >180 mmHg] and diastolic [<60 mmHg and >100 mmHg].

#### • Heart Rate:

Normal parameters: HR detection between 60-100 bpm.

Red Alert: Detection of HR < 50 bpm outside sleep period; or HR > 100 bpm (concurrently assessed by watch)

#### Oxygen Saturation:

Normal parameters: 95 – 100%

Yellow Alert: 91 – 95%

Red Alert: <90%

The conduct and actions planned to be taken by the clinical team after receiving the alerts through the Si3 platform (on D+1), as well as the guidelines that teleassisted patients will receive at the time of hospital discharge, are described in the table below:









#### INFORMAÇÕES À EQUIPE CLÍNICA

| | SITUAÇÃO | ORIENTAÇÃO | INTERVENÇÃO | AÇÃO |
|---|---|---|---|---|
| | Detecção de FC < 50 bpm fora do período de sono | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira<br>da equipe pelo telefone | Analisar os parâmetros clínicos e os sintomas do paciente. Enfermeira aciona teleconsulta com o médico se necessário. Em caso de necessidade, o médico orienta o paciente a procurar o PS do InCor |
| | Deteção de FC > 100 | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira informando o ocorrido | Orienta o paciente a procuraro PS do InCor |
| | PAS: Sistólica < 90 e > 180 mmHg | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | | Orienta o paciente a procurar o PS do InCor |
| | PAS: Diastólica < 60 e > 110 mmHg | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | - | Orienta o paciente a procurar o PS do InCor |
| | PAS: Sistólica 140 - 180 mmHg | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira<br>da equipe pelo telefone | Analisar os parâmetros clínicos e os sintomas do paciente. Enfermeira aciona teleconsulta com o médico se necessário. Em caso de necessidade, o médico orienta o paciente a procurar o PS do InCor |
| | PAS: Diastólica 90 - 110 mmHg | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira<br>da equipe pelo telefone | Analisar os parâmetros clínicos e os sintomas do paciente. Enfermeira aciona teleconsulta com o médico se necessário. Em caso de necessidade, o médico orienta o paciente a procurar o PS do InCor |
| • | SPO <sup>2</sup> : 91 - 95% | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira<br>da equipe pelo telefone | Analisar os parâmetros clínicos e os sintomas do paciente. Enfermeira aciona teleconsulta com o médico se necessário. Em caso de necessidade, o médico orienta o paciente a procurar o PS do InCor |
| | SPO <sup>2</sup> : <90% | Realizar medidas de parâmetros<br>indiretos (ECG, P.A. E SPO²) | Entrar em contato com a enfermeira da equipe pelo telefone | Orienta o paciente a procurar o PS do InCor |
| | Sono: < 7 horas contínuas | N/A | Entrar em contato com a enfermeira da equipe pelo telefone | Analisa a possível causa e fornece orientação de<br>Higiene do Sono |
| | Passos: <500 passos | N/A | Entrar em contato com a enfermeira da equipe pelo telefone | Analisa a possível causa e orienta o paciente a aumentar o nº de passos |

 Table 2. Flow of care for patients in the study (alerts, guidelines, interventions and actions)



The institutional electronic medical record (Si3) software modeling that will be used in the project to access clinical and functional information regarding patient data, are exemplified in the figures below:



Figure 6. Institutional Electronic Health Record: Macro view of the alerts referring to the teleassisted group.











Figure 7. Institutional Electronic Medical Record: Macro view of the alerts referring to each patient that makes up the teleassisted group.



Figure 8. Institutional Electronic Medical Record: Visualization of alerts referring to the variable and to each patient that makes up the teleassisted group.







#### 3.1 2 Ethical Aspects

The researcher in charge will ensure that obtaining the TCLE (Annex 1) is conducted in accordance with the specifications and international regulatory requirements of the ICH (International *Council for Humanization of Technical Requirements for Pharmaceuticals for Human Use*) for good clinical practices based on the ethical principles established by the resolution of the National Health Council (CNS, Resolution nº 466/2012).

be submitted to the CAPPesq Research Ethics Committee, via Plataforma Brasil. The ethical aspects of research involving human beings will be considered, as recommended by Resolution 466/2012. All data collected from volunteers will be treated ensuring confidentiality and meeting the other requirements established by the LGPD. The patients will be monitored by the multidisciplinary team via SI3, and any intercurrence verified by the multidisciplinary team in a "near real time" period and the patient will be consulted and guided in the face of the detected intercurrences.

After completing the survey, the data will be anonymized and analyzed by the InCor team. The raw data will be made available to the contracting company without any identification of the patient. After processing and analyzing the data, publication of the results in scientific databases is expected.





#### 4. ESTIMATED SCHEDULE

| ACTIVITIES | 1st<br>month | 2nd<br>month | 3rd-7th<br>month | 8th<br>month | 9th<br>month | 10th-<br>12th<br>month |
|---|---|---|---|---|---|---|
| Clinical PT submission to<br>the Scientific Committee<br>and CAPPesq | х | | | | | |
| Analysis of the Clinical PT<br>by the Research Ethics<br>Committee | х | х | | | | |
| Device Software<br>Installation and Testing | | | х | | | |
| Execution of the Clinical Protocol (inclusion of patients and remote monitoring) | | | х | | | |
| Compilation and analysis of results | | | | х | | |
| Final report | | | | х | х | |
| Accountability | | | | | x | |
| Submission of scientific articles | | | | | | х |





#### 5. ANNEXES

### 5.1. Case Report Form (CRF)

**CLINICAL TRIAL/UNIT: INOVA InCor** 

PRINCIPAL INVESTIGATOR: Dr. Fabio Biscegli Jatene

#### **CASE REPORT FORM**

#### **Study Title**

Wearable -assisted digital telemonitoring of post-cardiovascular surgery patients

#### **Study Samsung FAPO-x**

| EXECUTING RESEARCHER: Dr | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| I am confident that the infor<br>accurate. I confirm that the | | | | | | | | | | | | |
| changes to the protocol and | that t | writt | en in | forme | ed co | nsent | was | obtai | ned p | rior t | o the | study |
| Investigator Signature: | | | | | | | | | | | | |
| invostigator orginature. | | | | | | | | | | - | | |
| | | | Pati | ent N | lame | | | | | | | |
| | | | | | | | | | | | - | |
| Patient Signature: | | | | | | | | | | | | |
| | | _ | | | | | | | | | | |
| Signing date: | | | | | | | | | | ] | | |
| | D | d | m | m | m | Th | Th | Th | Th | | | |





| Inc | lusion criteria | Yes | No |
|---|---|---|---|
| 1 | Is the subject older than 22 years old with heart disease? | | |
| 2 | Did the subject voluntarily give written informed consent? | | |
| 3 | Does the subject agree to adhere to the study procedures? | | |
| 4 | Does the subject have surgical indication in the presence of heart disease? | | |
| 5 | | | |
| *If a | any inclusion criteria is marked as no, the patient is not eligible for the dy. | | |
| Ex | clusion criteria | Yes* | No |
| 1<br>1 | Did the subject have post-surgical complications with an extension of the hospital stay for more than 14 days? | Yes* | No |
| | Did the subject have post-surgical complications with an extension of | Yes* | No |
| 1 | Did the subject have post-surgical complications with an extension of the hospital stay for more than 14 days? Does the subject have any skin pathology or skin diseases? ( ex : | Yes* | No |
| 1 | Did the subject have post-surgical complications with an extension of the hospital stay for more than 14 days? Does the subject have any skin pathology or skin diseases? (ex: vitiligo, lupus and/or atopic dermatitis) Does the subject have allergies to the material components of the | Yes* | No |
| 1 2 3 | Did the subject have post-surgical complications with an extension of the hospital stay for more than 14 days? Does the subject have any skin pathology or skin diseases? (ex: vitiligo, lupus and/or atopic dermatitis) Does the subject have allergies to the material components of the mobile device? | Yes* | No |







## **VISIT 1 (TRIAGE)**

| | Date: |
|---|---|
| INFORMED CONSENT | |
| Note: Written informed consent must be given before a any current therapy is discontinued for the purposes of | |
| Did the subject freely give written informed consent? | Yes No |
| DEMOGRAPHIC DATA | |
| Age years): Fri: F | Teminine Masculine |
| Height (m): | • |
| Weight (Kg): | |
| BMI (BMI = Weight ÷ (Height × Height)): | |
| Race: | |
| Education Grade: | |
| CLINICAL EVALUATION: | |
| ( ) Altered heart rhythm ( ) Signs of HF ( ) Dizziness/fed | eling faint |
| ( ) Decrease in exercise tolerance, dyspnea ( ) Transie | nt Ischemic Attack |
| ( ) Stroke ( ) Chest pain ( ) Dyspnea at rest | |
| ( ) Exercise intolerance | |
| Da | te of Symptom Onset: |
| other, please specify | |







| COMBITIES: |
|---|
| ( ) Valvular Heart Disorder ( ) Diabetes Mellitus ( ) Hypertension |
| () COPD () Hyperthyroidism () TIA/CVA (history) |
| ( ) Sudden cardiac death in FH |
| PREVIOUS PROCEDURES: |
| () No Procedures |
| ( ) Coronary Angioplasty ( ) Revascularization Surgery ( ) Pacemaker |
| ( ) Cardiac Resynchronization Therapy ( ) Valve Prosthesis |
| ( ) Implantable cardiodefibrillator ( ) Ventricular Assist Device |
| ( ) Heart Transplantation ( ) Chemical Cardioversion ( ) Electrical Cardioversion |
| () Float Transplantation () Onemical Garacteristic () Electrical Garacteristic |
| SMOKING: |
| Yes No |
| TesNO |
| ( ) Current (Consumer for a period not less than 6 months) ( ) Past (If you have smoked at some point in your life, but have not smoked for more than 6 months) |
| DRINKING: |
| Yes No |
| ( ) Current (Consumer for a period not less than 6 months) ( ) Past (If you have smoked at some point in your life, but have not smoked for more than 6 months) |
| The report or record of consumption of alcoholic beverages, alcoholism and/or alcohol intoxication will be considered in this study. According to the World Health Organization (WHO) acceptable consumption is up to: 15 drinks/week for men and 10 drinks/week for women |







| ILLIC | CIT DRUGS : | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | Yes No | | 7 |
| Snoo | if | | | | | | | _ |
| Spec | | | | | | - | | |
| PHYS | SICAL EXERCISE: | | | | | | | |
| | SIGAL EXERCICE. | | | | | | | |
| | | | | | | Yes No | | |
| Spec | ifv· | | | | | | | |
| | ···y· | | | | | - | | |
| INGE | STION OF MEDICIN | IES | | | | | | |
| | subject currently or prements? | eviously | y taking | g any m | edicatio | ons, including vitamins and | d/or | |
| '' | | | | | | Yes No | | |
| * Rec | ord <b>all</b> medications on | the Co | ncomit | ant Med | dications | s page | | _ |
| MEDI | CAL HISTORY | | | | | | | |
| Is the | re any relevant medic | al histo | ory on | the foll | owing | systems? | _ | |
| Code | System | *Yes | No | | Code | System | *Yes | No |
| 1 | Cardiovascular | | | | 9 | neoplasm | | |
| two | Respiratory | | | | 10 | Neurological | | |
| 3 | Hepatobiliary | | | | 11 | Psychological | | |
| 4 | Gastrointestinal | | | | 12 | Immunological | | |
| 5 | genito-urinary | | | | 13 | Dermatology | | |
| 6 | Endocrine | | | | 14 | allergies | | |
| 7 | Hematological | | | | 15 | Eyes, ear, nose, throat | | |
| a | Skeletal muscle | 1 | 1 | 1 | 00 | Other | | |

<sup>\*</sup> If **YES** to any of the above, please enter the code for each condition in the boxes below, provide further details (including dates) and indicate whether the condition is







currently or potentially active. If providing details of surgery, specify underlying cause. Use a separate line for each condition.

| | Curren | | | |
|---|---|---|---|---|
| Code | Details (including dates) | | Yes | No |
| PHYSIC | AL EXAMINATION (To be performed only by the med | lical team) | | |
| Code | System | *Not<br>normal | Nor | mal |
| 1 | General appearance | | | |
| two | Cardiovascular | | | |
| 3 | Respiratory | | | |
| 4 | Gastrointestinal / Abdomen | | | |
| 5 | extremities | | | |
| | <b>ORMAL</b> , enter the code for each condition in the boxes belo se one _ line separate for each condition . | w and provic | le brief | detail |
| Code | Details | | | |
| VITAL S | SIGNS | | | |
| Pulse | bpm | | | |
| Pressure sitting) | Sanguine ( / mmHg | | | |







| ECG | Normal Not normal | *: | k | |
|---|---|---|---|---|
| | ( ) Sinus ( ) Atrial Fibrillation ( ) Atrial Flutter ( ) Nodal or Atrioventricular Reentry Tachycardia ( ) Wide QRS Tachycardia ( ) Bradyarrhythmias | | | |
| Store | Store the signed and dated dash in the plastic sleeve on the back of the CRF | | | |
| LAB | ORATORY ANALYSIS | | | Initials |
| Blood | Blood for hematology and biochemistry harvested by | | | |
| ✓ | ✓ Collection Date ( dd mmm yyyy ) | | | |
| | Hematology | | | |
| | Biochemistry | | | |

Please insert a copy of all results in the plastic sleeve on the back of the CRF.

#### **CONCOMITANT MEDICATION**

| Medication | Daily<br>Dose<br>(total) | Items | Reason | Start date<br>(MM/DD/YYYY) | End Date<br>(MM/DD/YYYY) | Continuous |
|---|---|---|---|---|---|---|
| | | | | / | / | |
| | | | | / | / | |
| | | | | / | / | |
| | | | | / | / | |
| | | | | / | / | |
| | | | | / | / | |
| | | | | / | / | |







| | | | | / | / |
|----------------------|------------------|----|----|---|---|
| | | | | / | / |
| Study End<br>(MM/DD/ | d Date:<br>YYYY) | /_ | /. | | |

### STUDY CLOSURE FORM

| Reason for Terminating Study (Please tick main reason only. Reasons other than Completed Study require explanation next to answer) Study Concluded Adverse Event/Severe Adverse Event (complete the Adverse Event form, if applicable) |
|---|
| Lost to follow |
| Participant no compatible |
| Medication Concurrent |
| Medication Contraindicated |
| To remove consent |
| Death |
| Other |







#### 5. 2. Term of Loan Responsibility





| l, | | | | , | bearer | of | RG |
|---|---|---|---|---|---|---|---|
| No | | UF, | resident | and | domici | led | at |
| Address | 3 | | | , | | | |
| No | Bairro | , City_ | | , | State | | Tel. |
| With.: _ | | , Tel. Answer: | | <u>-</u> | | | |

I inform, for the due purposes, that I received from INSTITUTO DO CORAÇÃO/FUNDAÇÃO ZERBINI registered with CNPJ under no. 50.644.053/0001-13, the equipment described below, owned by SAMSUNG ELETRÔNICA DA AMAZÔNIA LTDA., registered with CNPJ 23.209.756/0001-40, for exclusive use in the FAPO-X Samsung project of InovalnCor - InCor, for the term from 30 to 33 day(s) from this date, committing myself to return it in perfect condition at the end of this period.

I declare responsibility for their conservation, in accordance with the manufacturer's recommendations; committing myself not to lend or entrust to another person; and communicate, immediately to the **InovalnCor** via message to us **nº 11 XXXXXXXX, 11 XXXXXXXX** any incident and occurrence with the equipment(s); as well as ensuring the necessary precautions for the proper functioning and integrity of the assigned equipment, it being important to point out that the change of address (equipment) is not authorized without the knowledge and authorization of Inova InCor.

At the end of the monitoring period or, in case of withdrawal from the project, I will return the complete equipment and in perfect condition, considering the time of use, to the competent sector.

| Gadgets | Model | Accessories | Serial number |
|---------------------|-------|-----------------------|---------------|
| Smartwatch galaxy 5 | | Induction Charger | |
| smartphone | | USB Cable + Power Sup | |







| São Paulo, of | of 20 |
|---------------------|------------------|
| Studies Coordinator | Research Subject |





## 5.3. Activity Diary

| | Notes until lunch | | |
|------|-------------------|----------|-----------|
| Hour | Activities | Symptoms | Medicines |

| | Notes after lunch until dinner | | |
|------|--------------------------------|----------|-----------|
| Hour | Activities | Symptoms | Medicines |

| | Notes after dinner (don't forget times you slept and woke up) | | |
|---|---|---|---|
| Hour | Activities | Symptoms | Medicines |

| Time you slept: 1 | Гіте you woke up: |
|-------------------|-------------------|
|-------------------|-------------------|

| Date | Hour | Symptoms (palpitations, chest pains, fainting, dizziness, vertigo, etc. ) | Comments |
|---|---|---|---|







| Blood Pressure Monitoring | | | | | |
|---------------------------|------|-----|------|-----------|---------|
| Date | Hour | max | mine | Frequency | Therapy |





#### 6. REFERENCES

- <sup>1</sup> Malta DC, Bernal RTI, Lima MG, Araújo SSC, Silva MMA, Freitas MIF et al. Chronic non-communicable diseases and the use of health services: analysis of the National Health Survey in Brazil. Rev. Public Health . 2017; 51( Suppl 1): 4s.
- <sup>2</sup> Polanczyk CA. Epidemiology of cardiovascular diseases in Brazil: the truth hidden in the numbers. Arch bras Cardiol . 2020; 115(2):161-2.
- <sup>3</sup>Oliveira GMM, Brant LCC, Polanczyk CA, Biolo A, Nascimento BR, MDC et al. Cardiovascular Statistics Brazil 2020. Arq. Bras. Cardiol . 2020; 115(3): 308-439.
- <sup>4</sup>Feitosa ACR, Marques AC, Caramelli B, Ayub B, Polanczyk CA., Jardim C et al. II Guideline for Perioperative Assessment of the Brazilian Society of Cardiology. Arch. Bras. Cardiol.2011; 96 (3 Suppl 1): 1-68.
- <sup>5</sup>Stevens B, Pezzullo L, Verdian L, Tomlinson J, George A, Bacal F. The Costs of Heart Disease in Brazil. Arch . Bras. Cardiol . 2018; 111(1): 29-36.
- <sup>6</sup>The International Surgical Outcomes Study group. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries.British Journal of Anesthesia . 2016; 117(5): 601-609.
- <sup>7</sup> Michael F. Innovations in monitoring from smartphones to wearables. ICU Management & Practice 3 2017;148-50
- <sup>8</sup>da Silva PLN, Damasceno RF. Nosocomial infections in patients undergoing cardiac surgery: a review of incidences regarding post-surgery risk factors. J Manag Prim Health Care . 2020; 12:1-23.
- <sup>9</sup> Baeza-Herrera LA, Rojas-Velasco G, Márquez-Murillo MF, Portillo-Romero ADR, Medina-Paz L, Álvarez-Álvarez R et al. Atrial fibrillation in cardiac surgery. Arch Cardiol Mex. 2019;89(4):348-359.
- <sup>10</sup> Filardo G, Damiano RJ, Ailawadi G, Thourani VH, Pollock BD, Sass DM, et al. Epidemiology of new-onset atrial fibrillation following coronary artery bypass graft surgery. Heart. 2018;104(12):985–92.
- <sup>11</sup> Ronsoni RM, Souza AZM, Leiria TLL, Lima GG. Update on management of postoperative atrial fibrillation after cardiac surgery. Braz J Cardiovasc Surg 2020;35(2):206-10.
- <sup>12</sup> Goyal, P., Kim, M., Krishnan, U., Mccullough, SA, Cheung, JW, Kim, LK, ... & Kamel, H. (2022). Post-operative atrial fibrillation and risk of heart failure hospitalization. European heart journal, 43(31), 2971-2980.





- <sup>13</sup> A lTurki, A., Marafi, M., Proietti, R., Cardinale, D., Blackwell, R., Dorian, P., ... & Huynh, T. (2020). Major adverse cardiovascular events associated with postoperative atrial fibrillation after noncardiac surgery: a systematic review and meta-analysis. Circulation: Arrhythmia and Electrophysiology, 13(1), e007437.
- <sup>14</sup> Chon, KH, & McManus, DD (2018). Detection of atrial fibrillation using a smartwatch. Nature Reviews Cardiology, 15(11), 657-658.
- <sup>15</sup> Verzani RH, Serapiao ABS. Technological contributions to health: look at physical activity. Science health collective . 2020; 25(8): 3227-3238.
- <sup>16</sup> Businesswire . UCSF and Sage Bionetworks Announce Stress Research Study Leveraging New Sensor Technologies on the Samsung Galaxy S9 ans S9+. <a href="https://www.businesswire.com/news/home/20180315005916/en/UCSF-Sag">https://www.businesswire.com/news/home/20180315005916/en/UCSF-Sag</a>
- <sup>17</sup> Baig MM, Gholam HH, Moqeem AA, Mirza F, Linden MA. Systematic Review of Wearable Patient Monitoring Systems Current Challenges and Opportunities for Clinical Adoption. J Med Syst 2017; 41:115.
- <sup>18</sup>Dias D, Paulo Silva Cunha J. Wearable Health Devices-Vital Sign Monitoring, Systems and Technologies. Sensors (Basel). 2018;18(8):2414.
- <sup>19</sup> Subbe CP, Duller B, Bellomo R. Effect of an automated notification system for deteriorating ward patients on clinical outcomes. Crit Care. 2017 Mar 14;21(1):52.
- <sup>20</sup>Bove LA. Increasing Patient Engagement Through the Use of Wearable Technology. Journal for Nurse Practitioners. 2019; 15:535-9.
- <sup>21</sup> Bayoumy K, Gaber M, Elshafeey A et al. Smart wearable devices in cardiovascular care: where we are and how to move forward. Nat Rev Cardiol (2021).
- <sup>22</sup>Kolovos P. Wearable Technologies in Post-Operative Recovery: Clinical Applications and Positive Impacts. Intl J Caring Sciences. 2020;13(2):1474. <sup>23</sup>GFK. The technologies shaping consumers' lives now and next. Report GfK: Tech Trends 2017.
- <sup>24</sup>Slade SJA, Veillette CJ. The application of wearable technology in surgery: ensuring the positive impact of the wearable revolution on surgical patients. Front Surg. 2014; 1:39.
- <sup>25</sup>Adler-Milstein, J., Holmgren, AJ, Kralovec, P., Worzala, C., Searcy, T., & Patel, V. (2017). Electronic health record adoption in US hospitals: the emergence of a digital "advanced use" divide. Journal of the American Medical Informatics Association, 24(6), 1142-1148.
- <sup>26</sup> Vuppalapati, C., Ilapakurti, A., & Kedari, S. (2016, March). The role of big data in creating sense ehr, an integrated approach to creating next generation mobile sensor and wearable data driven electronic health record (ehr). In 2016







IEEE second international conference on big data computing service and applications (BigDataService) (pp. 293-296). IEEE.

- <sup>27</sup>Sutton, RT, Pincock, D., Baumgart, DC, Sadowski, DC, Fedorak, RN, & Kroeker, KI (2020). An overview of clinical decision support systems: benefits, risks, and strategies for success. NPJ digital medicine, 3(1), 1-10.
- <sup>28</sup> Alcade PR, Kirsztajn GM. Expenditures of the Brazilian Unified Health System with Chronic Kidney Disease . Braz. J. Nephrol . 2018;40(2):122-129
- <sup>29</sup>Bittar OJN, Biczyk M, Serinolli MI, Novaretti MCZ, Moura MMN. Health information systems and their complexity. Rev ADM in Health. 2018; 18:70. <sup>30</sup>Gutierrez MA, Rabelo MFS, Silva UTA, Furuie SS, Pires FA. InCor's experience in Health Information Systems. Goldbook of the 50th HUPE Scientific Congress. 2012.
- <sup>31</sup> Harris, PA, Taylor, R., Thielke, R., Payne, J., Gonzalez, N., & Conde, JG (2009). Research electronic data capture (REDCap)—a metadata-driven methodology and workflow process for providing translational research informatics support. Journal of biomedical informatics, 42(2), 377-381.